CLINICAL TRIAL: NCT04206150
Title: The Appropriate Level of Continuous Adductor Canal Block in Patients Undergoing Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2019-1038
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Degenerative Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Ninety six patients scheduled for total knee arthroplasty will be randomly divided into the three groups. In group 1, the adductor canal catheter is inserted at femoral triangle apex (the proximal end of the adductor canal). In group 2, the adductor canal catheter is inserted femur length/15*2 cm above the location where the nerve block performed in group 1. In group 3, the adductor canal catheter is inserted femur length/15*2 cm below the location where the nerve block performed in group 1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1(femoral triangle apex) (Active Comparator): the adductor canal catheter is inserted at femoral triangle apex (the proximal end of the adductor canal)
  Interventions: Procedure: the three different sites of continous adductor canal block: the adductor canal catheter is inserted at femoral triangle apex
- Group 2(femur length/15*2 cm above) (Active Comparator): the adductor canal catheter is inserted femur length/15*2 cm above the location where the nerve block performed in group 1
  Interventions: Procedure: the three different sites of continous adductor canal block: the adductor canal catheter is inserted femur length/15*2 cm above the location
- Group 3(femur length/15 cm below) (Active Comparator): the adductor canal catheter is inserted femur length/15cm below the location where the nerve block performed in group 1.
  Interventions: Procedure: the three different sites of continous adductor canal block: the adductor canal catheter is inserted femur length/15 cm below the location

INTERVENTIONS:
Procedure: the three different sites of continous adductor canal block: the adductor canal catheter is inserted at femoral triangle apex — In group 1, the adductor canal catheter is inserted at femoral triangle apex (the proximal end of the adductor canal).
  Arms: Group 1(femoral triangle apex)
Procedure: the three different sites of continous adductor canal block: the adductor canal catheter is inserted femur length/15*2 cm above the location — In group 2, the adductor canal catheter is inserted femur length/15*2 cm above the location where the nerve block performed in group 1.
  Arms: Group 2(femur length/15*2 cm above)
Procedure: the three different sites of continous adductor canal block: the adductor canal catheter is inserted femur length/15 cm below the location — In group 3, the adductor canal catheter is inserted femur length/15 cm below the location where the nerve block performed in group 1.
  Arms: Group 3(femur length/15 cm below)

SUMMARY:
Adductor canal catheters are being used to provide continuous postoperative analgesia after total knee arthroplasty surgery (TKA). There is much debate about where is the best position of continuous adductor canal block in patients undergoing TKA. Therefore, the investigators aim to compare the postoperative pain at three different level of continuous adductor canal block. Ninety six patients scheduled for total knee arthroplasty will be randomly divided into the three groups. In group 1, the adductor canal catheter is inserted at femoral triangle apex (the proximal end of the adductor canal). In group 2, the adductor canal catheter is inserted femur length/15*2 cm above the location where the nerve block performed in group 1. In group 3, the adductor canal catheter is inserted femur length/15cm below the location where the nerve block performed in group 1.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing total knee arthroplasty

Exclusion Criteria:

* 1. Patients who have infection or had surgery on the thigh
* 2. The subject is a foreigner or illiterate
* 3. Patients who have cognitive dysfunction

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Pain : Visual Analogue Scale (VAS) for pain | Baseline (Before surgery)
  The visual analog scale(VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain." (10). The ends are defined as the extreme limits of the parameter to be measured(symptom,pain,health) orientated from the left(0, worst) to the right(10, best).
Pain : Visual Analogue Scale (VAS) for pain | postoperative day 1
  The visual analog scale(VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain." (10). The ends are defined as the extreme limits of the parameter to be measured(symptom,pain,health) orientated from the left(0, worst) to the right(10, best).
Pain : Visual Analogue Scale (VAS) for pain | postoperative day 2
  The visual analog scale(VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain." (10). The ends are defined as the extreme limits of the parameter to be measured(symptom,pain,health) orientated from the left(0, worst) to the right(10, best).

SECONDARY OUTCOMES:
muscle strength | Baseline (Before surgery)
  Quadriceps strength of both legs was assessed by placing the dynamometer on the anterior of the ankle, between the malleoli.
muscle strength | postoperative day 1
  Quadriceps strength of both legs was assessed by placing the dynamometer on the anterior of the ankle, between the malleoli.
muscle strength | postoperative day 2
  Quadriceps strength of both legs was assessed by placing the dynamometer on the anterior of the ankle, between the malleoli.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chuan A, Lansdown A, Brick KL, Bourgeois AJG, Pencheva LB, Hue B, Goddard S, Lennon MJ, Walters A, Auyong D; Continuous Catheters in Adductor Canal versus Femoral Triangle (The CAFE study) investigators. Adductor canal versus femoral triangle anatomical locations for continuous catheter analgesia after total knee arthroplasty: a multicentre randomised controlled study. Br J Anaesth. 2019 Sep;123(3):360-367. doi: 10.1016/j.bja.2019.03.021. Epub 2019 May 2. PMID 31056239
- [Background] Sztain JF, Khatibi B, Monahan AM, Said ET, Abramson WB, Gabriel RA, Finneran JJ 4th, Bellars RH, Nguyen PL, Ball ST, Gonzales FB, Ahmed SS, Donohue MC, Padwal JA, Ilfeld BM. Proximal Versus Distal Continuous Adductor Canal Blocks: Does Varying Perineural Catheter Location Influence Analgesia? A Randomized, Subject-Masked, Controlled Clinical Trial. Anesth Analg. 2018 Jul;127(1):240-246. doi: 10.1213/ANE.0000000000003422. PMID 29750695
- [Derived] Lee B, Park SJ, Park KK, Kim HJ, Lee YS, Choi YS. Optimal location for continuous catheter analgesia among the femoral triangle, proximal, or distal adductor canal after total knee arthroplasty: a randomized double-blind controlled trial. Reg Anesth Pain Med. 2022 Jun;47(6):353-358. doi: 10.1136/rapm-2021-103284. Epub 2022 Feb 16. PMID 35173020